This document is the Statistical Analysis Plan for the study:

| REG-80-2015 | NCT03653312 | Neuromuscular Electrical Stimulation in |
|-------------|-------------|-----------------------------------------|
| | | Acute Ischemic Stroke (NESA) |

Date: 11.06.2020

# Statistical analysis plan

NESA - A randomized controlled trial of NeuroMuscular Electric Stimulation in patients with lower extremity paresis due to acute ischemic stroke

### Section 1: Administrative information

# Title & trial registration

• 1a: Neuromuscular Electrical Stimulation in Acute Ischemic Stroke (The NESA study)

NESA is a parallel group, superiority, randomised controlled trial (RCT) investigating if early NMES during exercise is superior to exercise alone in improving walking distance and speed, function and quality of life in patients (40–85 years of age) with acute ischemic stroke.

• 1b: Trial registration: ClinicalTrials.gov Identifier: NCT03653312 (originally registered 31.08.2018)

#### Version

2: Version 1.0. Date: 03.04.2020

#### Protocol version

• 3: This statistical analysis plan (SAP) has been written based on the revised protocol approved by the Regional Committees on Health Research Ethics for Region Zealand (SJ-444; 25.09.2015). This SAP adheres to the Guidelines for the content of statistical analysis plans in clinical trials (1). The SAP was made publicly available before finalizing the data collection at the primary endpoint and before any analysis is commenced.

# Revisions

4a: Revision history

4b: Justification for revision

4c: Timing of revision

| Protocol | Updated SAP | Section | Reason | Date changed |
|----------|-------------|---------|--------|--------------|
| version | version no. | number | | |
| | | changed | | |

# Roles and responsibility

5: Names, affiliations, and roles of SAP contributors

### Principal investigator:

Henriette Busk PT, MSc, PhD fellow.

# Senior investigator:

Troels Wienecke, MD, PhD, Clinical Associate Professor (principal supervisor)

### Other academic supervisors:

Søren Thorgaard Skou, PT, PhD, Professor (primary co-supervisor)

Gert Kwakkel PT, PhD, Professor

## Senior statistician:

Inge Petersen

# **Signatures**

6a: SAP author:

Date: 11.06.2020.

• 6b: Senior statistician signature: Mae

Date: 11.06.2020,

Date: 11.06.2020,

6c: Primary co-supervisor signature:

6d: Principal supervisor:

Date: 11.06.2020,

# **Section 2: Introduction**

# Background

7: Synopsis of trial background

# Background

Annually there are about 15,000 new cases of stroke in Denmark and the number is expected to rise with about 40% by 2035 due to the increasing population of elderly (2). Stroke is associated with the highest odds of reporting severe disability and more individual domains of disability compared with other conditions and therefore might be considered to be the most common cause of complex disability (3); stroke survivors represent the largest group of Danes receiving early retirement incapacity benefits (4). Optimising exercise rehabilitation to improve functionality for stroke survivors would thus be of great importance for the individual patient, their relatives, and society (4, 5). Therapists perform functional motor ability rehabilitation with stroke patients, and early and intensive exercise has shown faster remission and improved functionality in patients with stroke (6-10). Muscle strength for stroke patients can be increased by the assistance of NMES (11-16). To our knowledge the effect of NMES in addition to exercise in the acute phase after an ischemic stroke (<2 days) has never been studied.

This would be of great importance for future rehabilitation worldwide.

# **Objectives**

8: Description of specific objectives and hypotheses

The objective is to examine the added effect of NMES in addition to exercise in the acute phase after ischemic stroke in patients with paresis of the lower extremities. The primary endpoint is change in objectively-measured function at 90 days after ictus; secondary endpoints include self-reported quality of life, cognitive assessment, performance-based impairment and memory, and others at 90 days after ictus.

### Hypotheses

We hypothesize that patients randomized to early NMES during exercise will improve significantly more in objectively-measured function than patients randomised to only exercising until 90 days after ictus.

### Section 3: Study methods

### Trial design

9: Brief description of design

This is a RCT (1:1 ratio) conducted at the Department of Acute Neurology at Zealand University Hospital, Region Zealand, Denmark, with blinded evaluation of the effect parameters. Interventions will be delivered by trained physiotherapists. The intervention group receive exercise combined with NMES. The control group receive only exercise. Patient and physiotherapist blinding cannot be maintained due to muscle contractions from electric stimulation. Exercise begins no later than day 2 after ictus. The exercise starts at the acute ward during hospitalisation. After 2 days at the acute ward, some patients will be

transferred to either another neurological ward at another hospital in the region, or they will be sent home. Exercise is conducted on all weekdays for two weeks with a physiotherapist at either the ward, the ward at the other hospital or in the patients' home. Every training session lasts for 12 minutes, with one session per day. The stimulation will be given through external pads on the paretic limb during all exercise sessions. Effect parameters will be evaluated at baseline as well as on days 14 and 90 respectively in order to observe changes over time. Evaluation on day 90 is the primary follow-up, to assess any lasting effects of the intervention.

The primary endpoint is the between-group difference in change in 6 minutes walk test (6MWT) between the group randomised to exercise with NMES and the group randomised to exercise therapy alone from baseline to the 90 days post ictus follow-up.

#### Randomisation

#### 10: Randomisation details

A priori, a nurse independent from the study made a random distribution of the 50 participants. The allocation was stored in opaque sealed envelopes prepared by the nurse and after the distribution the envelopes were only accessible to the central study coordinator. The central study coordinator only opened the sealed envelopes after informed consent and baseline measures had been obtained.

### Sample size

# 11: Full sample size calculation

The study is powered to detect a difference in change of 34.4 points between the two groups in the primary outcome 6MWT from baseline to 90 days follow-up. A 34.4-meter difference in change between groups in 6MWT is considered clinically relevant (17). To detect the difference 21 patients in each of the intervention groups is needed (assuming a common SD of 38.7 (17), power=80%, alpha level=0.05). We planned to recruit a total of 50 patients to account for loss to follow-up (20%).

### Framework

12. Description of hypothesis testing framework

Both primary and secondary outcomes will be assessed using a superiority framework, expecting that patients undergoing intensive exercise with use of NMES in the acute phase of ischemic stroke will experience greater improvements in objectively-measured function than patients undergoing exercise alone.

## Statistical interim analysis and stopping rules

• 13: Specification of planned interim analysis and/or stopping rules

Not applicable.

# Timing of outcome assessments

# • 14: Details of timing of all analyses

The primary follow-up (90 days) will be conducted 90 days post ictus. Primary and secondary outcomes will be analysed collectively by the Principal Investigator under supervision and control from an independent statistician. Data from all follow-ups (baseline, 14 days and 90 days) will be included in this analysis. Outcomes presented under Primary or Secondary Outcome Measures at ClinicalTrials.gov (ID: NCT03653312) will be reported in the RCT report.

# 15: Timing of outcome assessments

Table 1 presents an overview of baseline characteristics and outcomes assessed and their timing.

| | <u>Baseline</u> | 14 days | 90 days |
|---|---|---|---|
| Baseline characteristics | | | |
| Age | X | | |
| Gender | X | | |
| SSS-Score | X | | |
| Height | X | | |
| Weight | Х | X | X |
| Favourite hand | Х | | |
| Smoking and years | Х | | |
| Weekly alcohol consumption | Х | | |
| Walking aids before<br>hospitalisation -indoors | X | | |
| Walking aids before<br>hospitalisation -outdoors | X | | |
| Residential circumstance | X | | |
| Stairs in the house | X | | |
| Force reduction | X | | |
| Social status | Х | | |
| Employment status | Х | | |
| Side of infarction | X | | |

| Smoking status | X | | |
|--------------------------------------------------|---|---|---|
| Co-morbidities know before<br>Hospitalisation | X | | |
| Co-morbidities identified during hospitalisation | Х | | |
| Earlier identified function-<br>limited diseases | X | | |
| Cognitive assessments | | | |
| Montreal Cognitive<br>Assessment | | Х | Х |
| Becks Depression Inventory | | X | Х |
| Patient reported outcomes | | | |
| EQ-5D-5L | | X | X |
| Physical performance tests | | | |
| 6MWT | Х | X | Х |
| 10 MWT | Х | X | Х |
| Sit to stand | Х | X | Х |
| Timed up and go | Х | X | Х |
| Guralnik | Х | X | Х |
| Fugl-Meyer UE motor part | X | X | X |
| Fugl-Meyer total UE score | Х | X | X |
| Adverse events | - | | |
| Patient-reported at<br>Follow-up | | X | X |
| Medical record review | | | X |

EQ-5D-5L = EuroQol Group 5-Dimension Self-Report Questionnaire, MoCA = Montreal Cognitive Assessment 6MWT = 6 Minutes Walk Test, 10 MWT = 10 Meter Walk Test

# Statistical principles

# Confidence intervals and p values

• 16: Level of statistical significance and confidence intervals

All statistical tests carried out to assess the between-group effects, will consist of two-sided tests with a 5% significance level (p=.05).

17: Adjustment for multiplicity

Since this study has one clearly defined primary outcome and all other outcomes serve as supportive outcomes, no adjustments for multiplicity are needed.

18: Confidence intervals

All confidence intervals presented will be 95% and two-sided.

# Adherence and protocol deviations

19a: Definition of adherence to the intervention

Poor compliance is defined as participating in less than 8 of the 10 exercise sessions (80%) in both the intervention and the control group. Compliance with the supervised exercise sessions will be registered by the physiotherapist delivering the interventions.

• 19b: Description of how adherence will be presented

Adherence will be presented as the number and percentage of patients who participate in 8 or more supervised exercise therapy sessions.

 $\bullet$   $\,$  19c & 19d: Definition of protocol deviations and how they will be reported

The following is defined as a major protocol deviation which may compromise the scientific value of the trial:

- More than 20% loss to follow-up
- Less than 50% participated in at least 8 of the supervised exercise therapy sessions.

All major protocol deviations will be reported in the primary report.

### Analysis population

20: Definition of analysis populations

In the primary analysis of the trial outcomes and the safety analysis (adverse events), all patients will be included according to the treatment they were randomised to receive, following the Intention-To-Treat (ITT) principle. This is the full analysis set, defined as an analysis set being as complete and as close to the ITT principle of including all randomised patients as possible (18). In addition, a secondary per protocol analysis will be performed. The per protocol population excludes patients with poor compliance (see 19a and 19b), and patients that withdrew their consent to participate.

### Trial population

# Screening data

21: Reporting of screening data

The duration of the recruitment period (start and end date) and the total number of subjects screened for eligibility throughout the recruitment period will be reported. See also item 23 & 24.

### Eligibility

22: Summary of eligibility criteria

### Inclusion criteria

- Adults aged 40 to 85 years diagnosed (CT/MRI or clinically diagnosed)
   with ischemic stroke within 2 days after debut.
- Leg paresis (muscle strength 2-4)
- Modified Ranking Scale (mRS) 0-1
- Cognitive capacity to participate in the study

### Exclusion criteria

- Pacemaker or other implanted electrical appliances
- Current or previous leg blood clot
- Absolutely absent sensitivity in affected extremity
- Pregnancy
- Depression (insufficient medical treatment)
- Anamnestic alcohol or drug abuse
- Untreated hypertension (BT> 150/90) at inclusion
- Functional limiting heart disease
- Epilepsy
- Dementia and/or malign diseases

### Recruitment and withdrawals

23 & 24: Information to be included in the CONSORT flow diagram

The CONSORT flow diagram (19) will consist of the following:

- All patients assessed for eligibility throughout the recruitment period
- All patients meeting one or more of the exclusion criteria, with reasons
- All patients eligible for inclusion in the trial
- All eligible patients not consenting, with reasons
- All patients randomised for both treatment arms
- All patients receiving and not receiving the allocated treatment for both treatment arms

- All patients with follow-up assessments at the 14 and 90 days post ictus follow-up<sup>1</sup>
- Withdrawals/lost to follow-up, with reasons, and timing for both treatment arms
- Patients included in the ITT and per protocol analyses for both treatment

<sup>1</sup>Patients with complete primary outcomes (6MWT) will be summarised at each follow-up for both treatment arms.

## Baseline patient characteristics

25a: List of baseline characteristics to be summarised

MOCK table 1 (below) presents an overview of baseline characteristics that will be presented in the primary report.

• 25b: Details on descriptive summary of baseline characteristics Categorical data will be summarised by numbers (%). Continuous data will be summarised by mean (SD) if data is normal and median (IQR) if data is skewed. No formal tests for significant differences between groups at baseline will be performed, as this is not recommended by CONSORT (19).

# Section 6: Analysis

# **Outcome definitions**

• 26: Specification of outcomes and timing
Table 1 presents an overview of outcomes assessed and their timing. MOCK table
2 and 3 illustrate how the results of the primary and secondary outcomes and
the safety analysis will be presented in the primary report.

### Analysis method

27: What analysis methods will be used

Outcomes presented under Primary or Secondary Outcome Measures at ClinicalTrials.gov (ID: NCT03653312) will be reported in the primary RCT report.

The primary endpoint i.e. between-group differences in change in the 6MWT from baseline to 90 days follow up will be analysed in repeated measures mixed effect model with subject being a random factor and visit (i.e. baseline, 14 days-and 90 days follow up) and interaction between visit and treatment arm (exercise with NMES or exercise alone) being fixed factors (20). A confidence interval not including 34.4 meters or more in the 6MWT will be interpreted as a lack of a clinically meaningful difference. Secondary outcomes will be analysed using the same model if appropriate. Model assumptions will be analysed for

normal distribution of residuals and if the assumption of normality is violated, confidence intervals will be estimated using Bootstrapping estimation methods. We will report estimated marginal means with p-values and 95% CI for superiority assessment.

The occurrence of adverse events (AE) will be compared between groups at the 90-days follow up using the appropriate method, if sufficient number of AE occurs the Poisson regression model with a robust error variance or similar.

## Missing data

28: Handling of missing data

No imputation methods will be applied, as a repeated measures mixed model do not require complete cases (21).

### Additional analysis

29: Details of any additional analysis

No additional analyses are planned. However, if found relevant, secondary, exploratory analyses might be conducted.

#### Harms

30: Handling of adverse events

Non-serious adverse events (AE) and serious adverse events (SAE) are recorded by asking patients face to face at the follow-up assessments. Additionally, the medical records from the recruiting hospitals will be examined for all AEs occurring from inclusion until the 90 days post ictus follow-up. An AE is defined as any undesirable experience during follow-up leading to contact with the health care system (general practitioner or hospital). AEs will be analysed for AEs and SAEs separately. If an AE results in hospitalisation, prolonged inpatient hospital care, result in surgery, or if an AE is life-threatening, result in death, permanent disability or damage, they will be categorised as SAEs, according to the FDA definition (22). SAEs will include cardiovascular disease and stroke, gastrointestinal and pulmonary events, systemic and local infection (and treatment with antibiotics) and deep vein thrombosis, but also other AEs will be categorized as an SAE in accordance with the FDA definition above. For all AEs, date of health care system contact is noted. Furthermore, duration of SAEs and potential consequences of SAEs will be registered if possible. AEs and SAEs will be presented as illustrated in MOCK table 3.

#### Statistical software

31: Details of statistical package used for the analysis

The statistical analysis will be performed in R-studio version 1.1.264

# Operating procedures

# 32: Data management

The procedures for data collection and management was approved by the Danish Data Protection Agency (Region Zealand, REG-80-2015). Data entry and coding of the de-identified data will be conducted by trained staff. Personal information about patients is kept separate from the main data set and will not be shared with anyone outside the central study team. To protect confidentiality before, during and after the trial, all personal data is stored securely. This SAP will form the basis for all analyses of the primary and secondary endpoints, which will be carried out by the Principal Investigator without any involvement from the study chairs. An assistant not involved in the study will code the two treatment arms into 'Group A' and 'Group B' before analysing the data. This will help ensure that the statistical analyses will be performed blinded from treatment allocation.

To reduce risk of interpretation bias, blinded results from the statistical analyses (Group A vs. Group B) will be presented to all authors, who will agree on two alternative written interpretations, one where group A is exercise WITH NMES and one where Group A is Exercise WITHOUT NMES. After finalising the blinded interpretation, the assistant will unblind who is Group A and Group B (23).

### References

- 1. Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Dore C, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. Jama. 2017;318(23):2337-43.
- 2. Rothwell PM, Algra A, Amarenco P. Medical treatment in acute and long-term secondary prevention after transient ischaemic attack and ischaemic stroke. Lancet (London, England). 2011;377(9778):1681-92.
- 3. Adamson J, Beswick A, Ebrahim S. Is stroke the most common cause of disability? Journal of Stroke and Cerebrovascular Diseases. 2004;13(4):171-7.
- 4. Flachs EM EL, Koch MB, Ryd JT, Dibba E, Skov-Ettrup L, Juel K. Sygdomsbyrden i Danmark Sygdomme: Statens Institut for Folkesundhed; 2015

[Available from: https://www.sst.dk/da/sygdom-og-behandling/~/media/00C6825B11BD46F9B064536C6E7DFBA0.ashx.

- 5. Andersen GD, D. Forchhammer, H.B. Iversen, H. Apopleksi -sygdom, behandling og organisation: Munksgaard; 2012.
- 6. Horn SD, DeJong G, Smout RJ, Gassaway J, James R, Conroy B. Stroke Rehabilitation Patients, Practice, and Outcomes: Is Earlier and More Aggressive Therapy Better? Archives of physical medicine and rehabilitation. 2005;86(12, Supplement):101-14.
- 7. Cumming TB, Thrift AG, Collier JM, Churilov L, Dewey HM, Donnan GA, et al. Very Early Mobilization After Stroke Fast-Tracks Return to Walking: Further Results From the Phase II AVERT Randomized Controlled Trial. Stroke; a journal of cerebral circulation. 2011;42(1):153-8.
- 8. Bohannon RW. Muscle strength and muscle training after stroke. Journal of rehabilitation medicine. 2007;39(1):14-20.
- 9. Ada L, Dorsch S, Canning CG. Strengthening interventions increase strength and improve activity after stroke: a systematic review. The Australian journal of physiotherapy. 2006;52(4):241-8.
- 10. Pradon D, Roche N, Enette L, Zory R. Relationship between lower limb muscle strength and 6-minute walk test performance in stroke patients. Journal of rehabilitation medicine. 2013;45(1):105-8.
- 11. Bowman BR, Baker LL, Waters RL. Positional feedback and electrical stimulation: an automated treatment for the hemiplegic wrist. Archives of physical medicine and rehabilitation. 1979;60(11):497-502.
- 12. Powell J, Pandyan AD, Granat M, Cameron M, Stott DJ. Electrical stimulation of wrist extensors in poststroke hemiplegia. Stroke; a journal of cerebral circulation [Internet]. 1999; 30(7):[1384-9 pp.]. Available from: <a href="http://onlinelibrary.wiley.com/o/cochrane/clcentral/articles/866/CN-00164866/frame.html">http://onlinelibrary.wiley.com/o/cochrane/clcentral/articles/866/CN-00164866/frame.html</a>.
- 13. Winchester P, Montgomery J, Bowman B, Hislop H. Effects of feedback stimulation training and cyclical electrical stimulation on knee extension in hemiparetic patients. Physical therapy. 1983;63(7):1096-103.
- 14. Newsam CJ, Baker LL. Effect of an electric stimulation facilitation program on quadriceps motor unit recruitment after stroke. Archives of physical medicine and rehabilitation. 2004;85(12):2040-5.
- 15. Eng JJ, Dawson AS, Chu KS. Submaximal exercise in persons with stroke: test-retest reliability and concurrent validity with maximal oxygen consumption. Archives of physical medicine and rehabilitation. 2004;85(1):113-8.
- 16. Sanford J, Moreland J, Swanson LR, Stratford PW, Gowland C. Reliability of the Fugl-Meyer assessment for testing motor performance in patients following stroke. Physical therapy. 1993;73(7):447-54.
- 17. Tang A, Eng JJ, Rand D. Relationship between perceived and measured changes in walking after stroke. Journal of neurologic physical therapy: JNPT. 2012;36(3):115-21.
- 18. Agency EM. ICH Topic E9 -Statistical Principles for Clinical Trials 1998. 2020.
- 19. Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. International journal of surgery (London, England). 2011;9(8):672-7.

- 20. J T, L B, T H, J R, M W, M H. Different ways to estimate treatment effects in randomised controlled trials. Contemporary clinical trials communications. 2018;10:80-5.
- 21. Ranstam J, Turkiewicz A, Boonen S, Van Meirhaeghe J, Bastian L, Wardlaw D. Alternative analyses for handling incomplete follow-up in the intention-to-treat analysis: the randomized controlled trial of balloon kyphoplasty versus non-surgical care for vertebral compression fracture (FREE). BMC medical research methodology. 2012;12:35.
- 22. FDA. <a href="https://www.fda.gov/safety/reporting-serious-problems-fda/what-serious-adverse-event">https://www.fda.gov/safety/reporting-serious-problems-fda/what-serious-adverse-event</a>.

  https://www.fda.gov/safety/reporting-serious-problems-fda/what-serious-adverse-event.
- 23. Jarvinen TL, Sihvonen R, Bhandari M, Sprague S, Malmivaara A, Paavola M, et al. Blinded interpretation of study results can feasibly and effectively diminish interpretation bias. J Clin Epidemiol. 2014;67(7):769-72.

# Mock tables

# Mock Table 1. Baseline characteristics

| Baseline characteristics | Exercise and NMES | Exercise |
|---|---|---|
| Sex | | |
| Age (years) | | Marian Washington Baseline |
| Weight (kg) | | |
| Body Mass Index | | |
| Comorbidities | | |
| Earlier function-limited diseases | | |
| Weekly alcohol consumption | | |
| Smoking status | | |
| Smoking (package-years) | | |
| Walking aids prior hospitalisation | | |
| Current Walking aids | | |
| Side of infarction | | |
| Level of force reduction | | |
| Received thrombolysis | | |
| SSS-score | | |
| Fugl-Meyer UE Motor Part | | |
| Fugl-Meyer Total score UE | | |
| 6 MWT | | |
| 10 MWT | | |
| Timed up and go | | |
| Sit to stand | | |
| Guralnik | | |

| Statistical Analysis Plan –NESA | Version1.0 |
|----------------------------------|------------|
| MOCA | |
| Becks Inventory Depression Scale | |
| EQ-5D-5L | |

Statistical Analysis Plan -NESA

Version1.0

Mock Table 2. Outcome at 90 days

| | Total no. of | Wean score at | Mean score at | Mean | Mean | Between-Group | Between-Group |
|---|---|---|---|---|---|---|---|
| | assessments | 90 days in | 90 days in | improvement In | improvement | difference in | difference in |
| | (exercise and | Exercise and | Exercise only | exercise and | in Exercise | mean | mean |
| | NMES | NMES group | group (95% CI) | MNES group | Only-group | improvement | improvement |
| | group/Exercise | (12 %56) | | (95% CI) | (95% CI) | (crude) | (adjusted) <sup>2</sup> |
| | Only group)1 | | | | | (95% CI) | (95% CI) |
| Primary | | | | | | | |
| outcome | | | | | | | |
| 6 MWT | | | | | | | |
| Secondary | | | | | | | |
| Outcomes | | | | | | | |
| 10 MWT | | | | | | | |
| Sit to stand | | | | | | | |
| Timed up and | | | | | | | |
| go | | | | | | | |

Statistical Analysis Plan -NESA

Version 1.0

| | | | | + | - | | | - | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | - |
| | | | | | | | | | 1 |
| | | | | | | | | | 900 |
| | | | | | | | | | 100 |
| | | | | | | | | | 100 |
| | | | | | | | | | 4:000 |
| | | | | | | | | | > |
| | | | | | | | | | 307 1/8 2 |
| ш | | ш | | | - | | | | 30), 000 |
| Fugl-Meyer UE | Motor part | Fugl-Meyer UE | <u>_</u> K | Guralnik | CA | ks | Depression | QOL Score | There were 1200 (195 v 8), 195 V 10 v 9)) seasible concernants for each events (200 at becaline and 500 at 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| Fug | Mot | Fug | Total | Gur | MOCA | Becks | Dep | 8 | Tho |

1200 ((25 x 8)+ (25 X 10 x 2)) possible assessments for each group (200 at baseline, and 500 at 14 days and at 90 days)

<sup>&</sup>lt;sup>2</sup> The results will be adjusted for baseline imbalance